CLINICAL TRIAL: NCT04338256
Title: Wellness and Resilience for College and Beyond: A Quasi-Experimental Pilot Study Investigating a Dialectical Behavior Therapy Skills-Infused College Course
Brief Title: Mental Health Curriculum Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Citrone 33 Foundation (Unknown)
Responsible Party: Principal Investigator, Carla Chugani, Assistant Professor of Pediatrics, University of Pittsburgh
Other Study IDs: STUDY18120150
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Mental Health Issue
Keywords: Mental Health Education; Public Health; Dialectical Behavior Therapy; College Students
MeSH Terms: interventions — Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Students enrolled in the Wellness Course: Students in this group are enrolled in the Wellness Course for the Spring 2020 or Fall 2020 semesters
  Interventions: Behavioral: Wellness and Resilience for College and Beyond (Undergraduate College Course)
- Controls: Students in this group are enrolled at study sites during the Spring 2020 or Fall 2020 semesters, but are not enrolled in the Wellness Course

INTERVENTIONS:
Behavioral: Wellness and Resilience for College and Beyond (Undergraduate College Course) — The course, "Wellness and Resilience for College and Beyond" was originally developed by James Mazza, PhD and colleagues at the University of Washington as a 10-week course. The course developers adapted their course materials to fit the needs of a 16-week semester for the purpose of this study. The Wellness Course teaches students evidence-based skills for improving mental health from dialectical behavior therapy, acceptance and commitment therapy, and the field of positive psychology. Classes meet for 2.5 hours weekly with approximately half of class time spent on teaching new content (lecture) and the other half spent with students working in small groups on practice and discussion exercises.
  Groups: Students enrolled in the Wellness Course

SUMMARY:
The purpose of this study is to investigate the acceptability, appropriateness, feasibility, and preliminary effectiveness of a college course grounded in skills from dialectical behavior therapy (DBT) titled, "Wellness and Resilience for College and Beyond." The study takes place on 5 college campuses in Pennsylvania and West Virginia offering the Wellness Course during the 2020 calendar year (Spring and Fall 2020 semesters). The Wellness Course is an undergraduate college course that includes 14 two and a half hour long lessons, weekly homework assignments and tracking of skills use via a "diary card," and a cumulative final exam at the end of the semester. Students who choose to enroll in the wellness course are offered the opportunity to enroll in the study and a comparison sample of students not enrolled are recruited from each site.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate College Students
* Enrolled at one of the five study sites

Exclusion Criteria:

* Students who are not undergraduates
* Students who do not fall within the age limits for the study (age 18-24 year)
* Students who are not enrolled at one of the five study sites

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is undergraduate college students recruited from five college campuses in Pennsylvania and West Virginia.
Sampling Method: Non-Probability Sample
Enrollment: 295 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Acceptability of the Wellness Course: Acceptability of Intervention Measure (AIM) | End of semester timepoint (approximately 4 months after baseline)
  Acceptability of Intervention Measure (AIM) is a 4 item scale. Respondents provide ratings using Likert type ratings ranging from 1-5, where 1= completely disagree and 5=completely agree. The ratings are summed and the average is taken.
Appropriateness of the Wellness Course: Intervention Appropriateness Measure (IAM) | End of semester timepoint (approximately 4 months after baseline)
  Intervention Appropriateness Measure (IAM) is a 4 item scale. Respondents provide ratings using Likert type ratings ranging from 1-5, where 1= completely disagree and 5=completely agree. The ratings are summed and the average is taken.
Feasibility of the Wellness Course: Feasibility of Intervention Measure (FIM) | End of semester timepoint (approximately 4 months after baseline)
  Feasibility of Intervention Measure (FIM) is a 4 item scale. Respondents provide ratings using Likert type ratings ranging from 1-5, where 1= completely disagree and 5=completely agree. The ratings are summed and the average is taken.

SECONDARY OUTCOMES:
Change in Use of Adaptive Coping Skills from Baseline to End of Semester (approximately 4 months after baseline) | Baseline and end of semester (approximately 4 months after baseline)
  Dialectical Behavior Therapy Ways of Coping Checklist (DBT WCCL) - Adaptive Skills Use Subscale. The DBT WCCL is a 59 item scale for which respondents provide ratings of their coping skills use on a Likert type scale from 0-3, where 0=Never Used and 3=Regularly Used. The adaptive coping sub-scale includes 38 items which are summed and averaged.
Change in Use of Adaptive Coping Skills from End of Semester (approximately 4 months after baseline) to 3-Month Follow-up | End of semester (approximately 4 months after baseline) and 3-month follow-up
  Dialectical Behavior Therapy Ways of Coping Checklist (DBT WCCL) - Adaptive Skills Use Subscale. The DBT WCCL is a 59 item scale for which respondents provide ratings of their coping skills use on a Likert type scale from 0-3, where 0=Never Used and 3=Regularly Used. The adaptive coping sub-scale includes 38 items which are summed and averaged.
Change in Use of Adaptive Coping Skills from Baseline to 3-Month Follow-up | Baseline and 3-month follow-up
  Dialectical Behavior Therapy Ways of Coping Checklist (DBT WCCL) - Adaptive Skills Use Subscale. The DBT WCCL is a 59 item scale for which respondents provide ratings of their coping skills use on a Likert type scale from 0-3, where 0=Never Used and 3=Regularly Used. The adaptive coping sub-scale includes 38 items which are summed and averaged.
Change in Emotion Dysregulation from Baseline to End of Semester (approximately 4 months after baseline) | Baseline and end of semester (approximately 4 months after baseline)
  Difficulties in Emotion Regulation Scale - Short Form is an 18 item scale. Respondents provide ratings on the frequency with which they struggle with various facets of emotion regulation using a Likert type scale ranging from 1-5, where 1= Almost Never (0-10% of the time and 5=Almost Always (91-100% of the time). Scores are summed and the average is taken.
Change in Emotion Dysregulation from End of Semester to 3-month follow-up | End of semester (approximately 4 months after baseline) and 3-month follow-up
  Difficulties in Emotion Regulation Scale - Short Form is an 18 item scale. Respondents provide ratings on the frequency with which they struggle with various facets of emotion regulation using a Likert type scale ranging from 1-5, where 1= Almost Never (0-10% of the time and 5=Almost Always (91-100% of the time). Scores are summed and the average is taken.
Change in Emotion Dysregulation from Baseline to 3-month follow-up | Baseline and 3-month follow-up
  Difficulties in Emotion Regulation Scale - Short Form is an 18 item scale. Respondents provide ratings on the frequency with which they struggle with various facets of emotion regulation using a Likert type scale ranging from 1-5, where 1= Almost Never (0-10% of the time and 5=Almost Always (91-100% of the time). Scores are summed and the average is taken.
Percent of Subjects with Past-30 Day Suicide Ideation at Baseline | Baseline
  Suicide Behaviors Questionnaire - Revised Version is a 4 item scale which assesses suicidality using a range of response options specific to each item, with items indicating higher risk being given more points. Item 1 assesses for suicide ideation and in this study, this is treated as a dichotomous variable.
Percent of Subjects with Past-30 Day Suicide Ideation at End of Semester (approximately 4 months after baseline) | End of semester (approximately 4 months after baseline)
  Suicide Behaviors Questionnaire - Revised Version is a 4 item scale which assesses suicidality using a range of response options specific to each item, with items indicating higher risk being given more points. Item 1 assesses for suicide ideation and in this study, this is treated as a dichotomous variable.
Percent of Subjects with Past-30 Day Suicide Ideation at 3-month follow-up | 3-month follow-up
  Suicide Behaviors Questionnaire - Revised Version is a 4 item scale which assesses suicidality using a range of response options specific to each item, with items indicating higher risk being given more points. Item 1 assesses for suicide ideation and in this study, this is treated as a dichotomous variable.
Change in Past-30 Day Suicide Risk from Baseline to End of Semester (approximately 4 months after baseline) | Baseline and end of semester (approximately 4 months after baseline)
  Suicide Behaviors Questionnaire - Revised Version is a 4 item scale which assesses suicidality using a range of response options specific to each item, with items indicating higher risk being given more points. Scores on all 4 items can be summed. In college students a sum score of greater than or equal to 7 is associated with current suicide risk.
Change in Past-30 Day Suicide Risk from End of Semester (approximately 4 months after baseline) to 3-month follow-up | End of semester (approximately 4 months after baseline) and 3-month follow-up
  Suicide Behaviors Questionnaire - Revised Version is a 4 item scale which assesses suicidality using a range of response options specific to each item, with items indicating higher risk being given more points. Scores on all 4 items can be summed. In college students a sum score of greater than or equal to 7 is associated with current suicide risk.
Change in Past-30 Day Suicide Risk from Baseline to 3-month follow-up | Baseline and 3-month follow-up
  Suicide Behaviors Questionnaire - Revised Version is a 4 item scale which assesses suicidality using a range of response options specific to each item, with items indicating higher risk being given more points. Scores on all 4 items can be summed. In college students a sum score of greater than or equal to 7 is associated with current suicide risk.

CONTACTS AND LOCATIONS:
Overall Officials: Carla D Chugani, PhD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - University of Pittsburgh, Greensburg Campus, Greensburg, Pennsylvania
  - Carlow University, Pittsburgh, Pennsylvania
  - Carnegie Mellon University, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chugani CD, Fuhrman B, Abebe KZ, Talis J, Miller E, Coulter RWS. Wellness and resilience for college and beyond: protocol for a quasi-experimental pilot study investigating a dialectical behaviour therapy skill-infused college course. BMJ Open. 2020 Jun 21;10(6):e036833. doi: 10.1136/bmjopen-2020-036833. PMID 32565475